CLINICAL TRIAL: NCT04285853
Title: Are Opioids Needed: A Double-Blinded, Randomized Controlled Trial and Examination of Predictors of Opioid Use Following ACL Reconstruction
Brief Title: Are Opioids Needed After ACL Reconstruction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Orthopedic Research and Education Foundation (Other)
Responsible Party: Principal Investigator, John Xerogeanes, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00116728
Record Dates: First submitted 2020-02-24; First posted 2020-02-26 (Actual); Results first posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-09

CONDITIONS: Anterior Cruciate Ligament Rupture
Keywords: Opioids
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Oxycodone

STUDY DESIGN:
Intervention Model Description: Prospective, double-blind, randomized controlled clinical trial
Who Masked: Participant, Investigator
Masking Description: Both participants and PI (orthopaedic surgeon) will be blinded. Placebo pills will be closely matched to oxycodone pills, so patients will not know to which group they are allocated. The PI will be blinded to group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxycodone Arm (Experimental): Patients in this opioid group will receive 15 oral opioid tablets (5 mg oxycodone) Patients will also receive 8 "rescue" medications, in the Oxycodone arm will be placebo "rescue" medications.
  All participants will also receive the following as part of standard of care:
  1. Oral non-opioid (1000 mg acetaminophen), every 8 hours.
  2. Prescription of non-opioid non-steroidal anti-inflammatory medication (naproxen 500 mg) to be used 2x/day post-surgery.
  3. Standardized multimodal intra- and post-operative protocols, including an adductor canal peripheral nerve block.
  4. Intraoperative education on post-surgical pain management.
  Interventions: Drug: Oxycodone
- Placebo Arm (Placebo Comparator): Patients in placebo group will receive 15 placebo tablets. All patients will also receive 8 "rescue" medications: Patients who randomize to the non-opioid arm will receive 5mg oxycodone "rescue" tablets.
  All participants will also receive the following as part of standard of care:
  1. Oral non-opioid (1000 mg acetaminophen), every 8 hours.
  2. Prescription of non-opioid non-steroidal anti-inflammatory medication (naproxen 500 mg) to be used 2x/day post-surgery.
  3. Standardized multimodal intra- and post-operative protocols, including an adductor canal peripheral nerve block.
  4. Intraoperative education on post-surgical pain management.
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Oxycodone — 5 mg oxycodone pills every 4-6 hrs if pain level 7 or higher on Numeric rating scale 1-10
  Other Names: Xtampza ER, Oxaydo, Roxicodone, and Oxycontin
  Arms: Oxycodone Arm
Drug: Placebo oral tablet — Placebo tablets (both trial and "rescue") will be matched to size, shape, color, and texture of oxycodone tablets.
  Arms: Placebo Arm

SUMMARY:
As the public health sector continues to confront the opioid epidemic, orthopaedic surgeons must revisit pain management protocols to reduce unnecessary opioid prescriptions. The long-term goal is to reduce opioid use and residual opioids in circulation.

DETAILED DESCRIPTION:
As the public health sector continues to confront the opioid epidemic, orthopaedic surgeons must revisit pain management protocols to reduce unnecessary opioid prescriptions. The long-term goal is to reduce opioid use and residual opioids in circulation. The purposes are to 1) conduct a double-blinded randomized controlled trial to determine the effectiveness of opioid versus non-opioid medications on post-surgical pain, and 2) examine predictors of opioid usage in individuals following Anterior Cruciate ligament (ACL) reconstruction. Patients will use an innovative Smartphone application to track pain and medication usage. Additionally, patients will complete quality of life and pain catastrophizing questionnaires, as well as undergo pain threshold testing, to be used in a model to determine predictors of greater post-surgical opioid use. This study will provide information on non-opioid alternatives and specific predictors of post-surgical opioid use that can be used to develop prescribing protocols. These findings will help orthopaedic surgeons make informed decisions when tailoring individualized prescriptions for patients following ACL reconstruction. Importantly, findings will be readily translatable into research to reduce opioid use in other orthopaedic surgical cohorts as well. Our ultimate goal is to lessen the burden of the opioid epidemic on not only our orthopaedic patients, but also society, by minimizing the number of opioids left in circulation.

ELIGIBILITY:
Inclusion Criteria:

* Males and females
* Aged 14-40 years
* Scheduled for primary (Anterior cruciate ligament) ACL reconstruction using quadriceps tendon autograft.

Exclusion Criteria:

* Revision and/or contralateral ACL reconstruction procedures
* Allergies to local anesthetics
* Chronic pain medication use
* Weight <50 kg, local infections
* Known coagulopathies,
* Liver dysfunction or renal failure

Ages: 14 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 98 (Actual)
Dates: Start 2020-09-16 (Actual); Primary Completion 2022-09-19 (Actual); Study Completion 2022-09-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Xerogeanes, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - The Emory Clinic, Atlanta, Georgia
  - Emory clinic at Executive Park, Atlanta, Georgia
  - Emory Orthopedic and spine Hospital, Tucker, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Oxycodone Arm: Patients in this opioid group will receive 15 oral opioid tablets (5 mg oxycodone) Patients will also receive 8 "rescue" medications, in the Oxycodone arm will be placebo "rescue" medications.
  All participants will also receive the following as part of standard of care:
  1. Oral non-opioid (1000 mg acetaminophen), every 8 hours.
  2. Prescription of non-opioid non-steroidal anti-inflammatory medication (naproxen 500 mg) to be used 2x/day post-surgery.
  3. Standardized multimodal intra- and post-operative protocols, including an adductor canal peripheral nerve block.
  4. Intraoperative education on post-surgical pain management.
  Oxycodone: 5 mg oxycodone pills every 4-6 hrs if pain level 7 or higher on Numeric rating scale 1-10
- Placebo Arm: Patients in placebo group will receive 15 placebo tablets. All patients will also receive 8 "rescue" medications: Patients who randomize to the non-opioid arm will receive 5mg oxycodone "rescue" tablets.
  All participants will also receive the following as part of standard of care:
  1. Oral non-opioid (1000 mg acetaminophen), every 8 hours.
  2. Prescription of non-opioid non-steroidal anti-inflammatory medication (naproxen 500 mg) to be used 2x/day post-surgery.
  3. Standardized multimodal intra- and post-operative protocols, including an adductor canal peripheral nerve block.
  4. Intraoperative education on post-surgical pain management.
  Placebo oral tablet: Placebo tablets (both trial and "rescue") will be matched to size, shape, color, and texture of oxycodone tablets.
Period: Overall Study
Arm/Group | Oxycodone Arm | Placebo Arm
Started | 49 | 49
Completed | 39 | 44
Not Completed | 10 | 5
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Lost to Follow-up | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oxycodone Arm | Placebo Arm | Total
Number analyzed (Participants) | 49 | 49 | 98
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.6 (6.9) | 20.6 (5.7) | 21.6 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 22 | 48
  Male | 23 | 27 | 50
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 12 | 13
  Not Hispanic or Latino | 14 | 0 | 14
  Unknown or Not Reported | 34 | 37 | 71
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 4 | 6
  White | 14 | 8 | 22
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 29 | 33 | 62
Region of Enrollment [Number; unit: participants]
  United States | 49 | 49 | 98
Body mass index [Mean (Standard Deviation); unit: kg/m2] | 24.0 (3.7) | 23.6 (3.8) | 23.8 (3.7)
Smoking status [Count of Participants; unit: Participants]
  Not a smoker | 34 | 34 | 68
  Current Cigarette User | 2 | 0 | 2
  Former smoker | 1 | 0 | 1
  Unknown status | 12 | 15 | 27
Current use of alcohol [Count of Participants; unit: Participants]
  Yes | 13 | 8 | 21
  No | 14 | 18 | 32
  Did not provide an answer | 22 | 23 | 45
Currently on treatment for depression [Count of Participants; unit: Participants]
  Yes | 4 | 2 | 6
  No | 45 | 47 | 92
ADHD treatment [Count of Participants; unit: Participants]
  Yes | 3 | 2 | 5
  No | 46 | 47 | 93
Preoperative opioid use [Count of Participants; unit: Participants]
  Yes | 0 | 1 | 1
  No | 49 | 48 | 97

OUTCOME MEASURES:

1. Primary Outcome: Pain Level: Numeric Rating Scale
Description: Patients will record pain levels on Numeric Rating Scale 1-10, where 1 is minimal pain and 10 is associated with highest level of pain (worse outcome).
Time Frame: Postoperative days 0-6
Population: Number analyzed in one or more rows differs from overall number analyzed depending on the number of patients that were able to provide data about their level of pain.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Oxycodone Arm | Placebo Arm
Number analyzed (Participants) | 40 | 42
score on a scale
  Study Day 0: number analyzed (Participants) | 37 | 41
  Study Day 0 | 4.6 [3.9 to 5.2] | 4.5 [4.0 to 5.1]
  Study Day 1: number analyzed (Participants) | 39 | 42
  Study Day 1 | 4.7 [4.1 to 5.2] | 5.1 [4.5 to 5.6]
  Study Day 2 | 3.8 [3.2 to 4.3] | 3.8 [3.3 to 4.4]
  Study Day 3: number analyzed (Participants) | 40 | 41
  Study Day 3 | 3.0 [2.6 to 3.5] | 3.3 [2.8 to 3.9]
  Study Day 4: number analyzed (Participants) | 36 | 38
  Study Day 4 | 3.0 [2.4 to 3.5] | 3.0 [2.4 to 3.5]
  Study Day 5: number analyzed (Participants) | 35 | 36
  Study Day 5 | 2.6 [2.1 to 3.2] | 2.9 [2.4 to 3.5]
  Study Day 6: number analyzed (Participants) | 33 | 37
  Study Day 6 | 2.9 [1.8 to 4.0] | 2.8 [2.3 to 3.4]

2. Other Pre Specified Outcome: Change in Pain Threshold Testing
Description: will be conducted with digital pressure dolorimeter (Wagner Force One Model FDIX 50TM, Wagner Instruments). Pressure dolorimeters are devices that measure pressure/pain threshold. The device will be held perpendicular to the areas to be tested. The force will be increased at a constant rate of 1 kg/cm2. Patients will be instructed to express pain either by saying "ouch" or raising their hand when pain is felt. The force read on the digital dolorimeters will be recorded. This procedure will be repeated 3 times. Both right and left sides will be tested.
Time Frame: Postoperative days 0-6, 6 weeks post-surgery
Reporting Status: Not Posted

3. Other Pre Specified Outcome: Change in Pain Catastrophizing Scale (PCS)
Description: It will be determined with the Pain Catastrophizing Scale (PCS). Pain catastrophizing is described as "an exaggerated negative mental set brought to bear during actual or anticipated painful experience." In other words, it is a feeling of helplessness. The PCS is a 13-item questionnaire that inquires about thoughts and feelings a patient experiences when in pain. Responses are recorded on a 5-point Likert scale ("not at all" to "all the time"). A total score is yielded ranging from 0-52. Higher score is associated with worse outcome.
Time Frame: Postoperative days 0-6, 6 weeks post-surgery
Reporting Status: Not Posted

4. Other Pre Specified Outcome: Change in Quality of Life: Euro Quality of Life Index (Euro QoL 5-D 5-L) EQ-5D
Description: Quality of life will be measured with the instrument Euro Quality of Life Index (Euro QoL 5-D 5-L) EQ-5D is a standardized measure of health status that measures five dimensions, Mobility, Self-care, Daily activities, Pain/Discomfort, Anxiety/ Depression. Each dimension can be rated at five levels: from no problems to major problems. The five dimensions can be summed into a descriptive health state with 11111 representing no problems in any of the five health dimensions and 55555 indicating major problems in any of the five health dimensions.
Time Frame: Postoperative days 0-6, 6 weeks post-surgery
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 6 weeks post-operatively
Arm/Group | Oxycodone Arm | Placebo Arm
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 15/49 | 8/49
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oxycodone Arm (N=49) | Placebo Arm (N=49)
Euphoria (Psychiatric disorders) | 0 (0) | 1 (1)
Nausea and vomiting (Gastrointestinal disorders) | 5 (5) | 2 (2)
Constipation (Gastrointestinal disorders) | 10 (10) | 4 (4)
Other (General disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-04): https://cdn.clinicaltrials.gov/large-docs/53/NCT04285853/Prot_SAP_000.pdf